CLINICAL TRIAL: NCT00861783
Title: A Phase 1 Dose-Escalation Study of the Safety and Clinical Effects of ON 01910.Na in Combination With Either Irinotecan or Oxaliplatin in Patients With Hepatoma and Other Advanced Solid Tumors
Brief Title: Safety of ON 01910.Na and Irinotecan or ON 01910.Na and Oxaliplatin in Patients With Hepatoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-08
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Hepatoma; Advanced Solid Tumor
Keywords: oxaliplatin; diaminocyclohexane oxalatoplatinum; oxalatoplatin; oxalatoplatinum; Eloxatin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Irinotecan; ON 01910; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - irinotecan (Experimental): Note: As of Amendment 2 (March 2009), treatment in the irinotecan arm of the study (Group A) is closed to enrollment.
  Treatment with escalating doses of ON 01910.Na in combination with irinotecan.
  Interventions: Drug: irinotecan and ON 01910.Na
- Group B - oxaliplatin (Experimental): Treatment with escalating doses of ON 01910.Na in combination with oxaliplatin.
  Interventions: Drug: oxaliplatin and ON 01910.Na

INTERVENTIONS:
Drug: irinotecan and ON 01910.Na — ON 01910.Na will be administered by IV infusion over 24 hours once per week in a 6-week cycle (6 doses per cycle). The dose of ON 01910.Na will start at 250 mg/m2 and will proceed to higher levels based on safety of the combination regimen in the previous cohort.
  Irinotecan 180 mg/m2 will initially be administered by IV infusion over 90 minutes q2 weeks of a 6-week cycle (3 doses per cycle). Dose modifications due to toxicity will be instituted according to approved labelling.
  Other Names: camptothecin-11; irinotecan HCl; Camptosar; CPT-11; diaminocyclohexane oxalatoplatinum; rigosertib sodium
  Arms: Group A - irinotecan
Drug: oxaliplatin and ON 01910.Na — ON 01910.Na will be administered by IV infusion over 24 hours once per week in a 6-week cycle (6 doses per cycle). The dose of ON 01910.Na will start at 250 mg/m2 and will proceed to higher levels based on safety of the combination regimen in the previous cohort.
  Oxaliplatin 85 mg/m2 will initially be administered by IV infusion over 120 minutes every 2 weeks of a 6-week cycle (3 doses per cycle). Dose modifications due to toxicity will be instituted according to approved labeling.
  Other Names: Eloxatin; oxaloplatinum; oxalatoplatin; rigosertib sodium
  Arms: Group B - oxaliplatin

SUMMARY:
Studies done in the laboratory have demonstrated beneficial effects of ON 01910.Na, a new, unapproved drug, when it is used in combination either irinotecan and oxaliplatin, two approved, extensively used anti-cancer drugs. In these laboratory studies, mice implanted with cells (Bel-7402 cells) that came from a human tumor were used as a model of liver cancer. In mice that were not treated, the Bel-7402 cells formed very large tumors. In mice that were treated with ON 01910.Na, irinotecan or oxaliplatin alone, growth of tumors was reduced compared to the untreated group. When a combination of ON 01910.Na and irinotecan or of ON 01910.Na and oxaliplatin was used to treat the mice, tumor growth was completely inhibited. Another observation in these studies was that toxicity did not increase when the combinations were used. These results and similar results from other studies support the hypothesis that a combination of ON 01910.Na and irinotecan or of ON 01910.Na and oxaliplatin would be an effective and tolerable treatment for liver and other types of cancer.

The primary objective of this phase 1 study is to find out what doses of ON 01910.Na in combination with either irinotecan or oxaliplatin are safe and tolerable in patients with liver and other types of cancer.

DETAILED DESCRIPTION:
This is an open-label, 2-arm, dose-escalation combination-therapy study in which patients with hepatoma and other advanced malignancies will be assigned by the Investigator to dosing with either irinotecan plus ON 01910.Na (Group A), or oxaliplatin plus ON 01910.Na (Group B). Note: As of Amendment 2 of this protocol, treatment in the irinotecan arm of the study (Group A) is closed to enrollment and patients will be enrolled only in Group B, the oxaliplatin treatment arm. Patients will be enrolled in 1 of 4 Cohorts (4 sequential Cohorts in Group B) of 3 patients each. Up to 6 additional patients will be tested at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years of age with histologically or cytologically confirmed hepatoma and other solid tumors that are metastatic or progressive, for whom no standard therapy holds curative potential and for whom irinotecan or oxaliplatin are reasonable treatment options.
* Patients must have evaluable disease, either measurable on imaging or with informative tumor marker(s).
* Eastern Collaborative Oncology Group (ECOG) Performance Status of ≤2.
* Life expectancy >12 weeks.
* Any acute or chronic adverse effects of prior chemotherapy have resolved to <Grade 2 as determined by CTCAE v3 criteria.
* Existing or planned central venous access with a 2-channel infusion catheter system.
* Laboratory values meet the following criteria: Absolute neutrophil count ≥1,500 cells/µL; Platelets ≥100,000 cells/µL; Total bilirubin ≤1.5 times the upper limit of normal; AST (SGOT) ≤2.5 times the upper limit of normal; ALT (SGPT) ≤2.5 times the upper limit of normal; Serum creatinine ≤1.5 mg/dL or a measured creatinine clearance ≥50 mL/min; Negative βhCG test in women of childbearing potential (defined as women ≤50 years of age or history of amenorrhea for ≤12 months prior to study entry).
* Patients with primary liver cancer or hepatic metastasis are eligible to enroll, provided they meet the following: Total bilirubin is ≤2 mg/dL; AST and ALT are each ≤5 times the institutional upper limit of normal; Ascites, if present, is manageable with diuretic agents alone.
* If there is a history of treated brain metastases, these must have been clinically stable for ≥4 weeks prior to enrollment.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Severe liver dysfunction (Child-Pugh Class C or uncompensated Class B with persistent encephalopathy, persistent ascites, or prothrombin time >1.5 times the upper limit of normal) is present.
* Patients with a history of esophageal bleeding are excluded unless arices have been sclerosed or banded and bleeding episodes have not occurred during the prior 6 months.
* Contraindications, including known hypersensitivity, to the assigned chemotherapy agent (i.e., irinotecan or oxaliplatin).
* Prior receipt of ON 01910.Na or prior participation in this protocol.
* Use of any investigational agents within 4 weeks of study enrollment.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the Investigator.
* Patients with ascites requiring active medical management including paracentesis, peripheral bilateral edema or hyponatremia (defined as serum sodium value of <134 Meq/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 6 - 12 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 - 12 months
tumor measurement | 6 - 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Takao Ohnuma, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- [Background] Jimeno A, Chan A, Cusatis G, Zhang X, Wheelhouse J, Solomon A, Chan F, Zhao M, Cosenza SC, Ramana Reddy MV, Rudek MA, Kulesza P, Donehower RC, Reddy EP, Hidalgo M. Evaluation of the novel mitotic modulator ON 01910.Na in pancreatic cancer and preclinical development of an ex vivo predictive assay. Oncogene. 2009 Jan 29;28(4):610-8. doi: 10.1038/onc.2008.424. Epub 2008 Nov 24. PMID 19029951
- [Background] Jimeno A, Li J, Messersmith WA, Laheru D, Rudek MA, Maniar M, Hidalgo M, Baker SD, Donehower RC. Phase I study of ON 01910.Na, a novel modulator of the Polo-like kinase 1 pathway, in adult patients with solid tumors. J Clin Oncol. 2008 Dec 1;26(34):5504-10. doi: 10.1200/JCO.2008.17.9788. Epub 2008 Oct 27. PMID 18955447
- [Background] Reddy MV, Mallireddigari MR, Cosenza SC, Pallela VR, Iqbal NM, Robell KA, Kang AD, Reddy EP. Design, synthesis, and biological evaluation of (E)-styrylbenzylsulfones as novel anticancer agents. J Med Chem. 2008 Jan 10;51(1):86-100. doi: 10.1021/jm701077b. Epub 2007 Dec 19. PMID 18088089
- [Background] Gumireddy K, Reddy MV, Cosenza SC, Boominathan R, Baker SJ, Papathi N, Jiang J, Holland J, Reddy EP. ON01910, a non-ATP-competitive small molecule inhibitor of Plk1, is a potent anticancer agent. Cancer Cell. 2005 Mar;7(3):275-86. doi: 10.1016/j.ccr.2005.02.009. PMID 15766665
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.